CLINICAL TRIAL: NCT05279911
Title: Influence of Low-level Laser Therapy on Radiographic and Biochemical Profiles in Type II Controlled Diabetic Patients After Dental Implant Insertion: A Randomized Case Control Study
Brief Title: Effect of Low-level Laser Therapy on Type II Controlled Diabetic Patients After Dental Implant Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Collaborators: Misr International University (Other); Al-Azhar University (Other); Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Mohamed Moawed Ibrahim Ghoneim, PhD, Assistant professor of Oral and Maxillofacial Surgery, Sinai University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: FWA00025577
Record Dates: First submitted 2022-02-24; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); Low-level Laser Therapy; Bone Density Increased
Keywords: T2DM (Type 2 Diabetes Mellitus); Dental Implant insertion; Osteoprotegrin (OPG); Bone Density; Low-level laser therapy; LLLT
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Osteosclerosis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Study design: A randomized case control study. A total of 40 adult participants of both genders of at least 21 years old were included in the study. All participants were controlled T2DM patients for more than 2 years (diagnosed according to the American Diabetes Association criteria) [21]. Patients were able and willing to participate in the study. Patients were recruited from out-patient clinic of Oral Diagnosis at Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Egypt.
Who Masked: Investigator
Masking Description: Patients were included in the study after fulfilling all the eligibility criteria and signing the informed consent form for participation and permission to use obtained data or research purposes. Patients were randomly allocated according to the type of treatment (control group: conventional implant placement and intervention group: LLLT) that were performed considering the implant as a unit. To ensure concealment of randomization, consecutively numbered envelopes were used. The team of surgeons only became aware of the type of intervention at the time of surgery, when the envelope was opened by a blinded investigator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Implants were randomly inserted in 20 non-lased T2DM patients (Control)
- Low level laser therapy (Experimental): Implant were randomly inserted in 20 lased T2DM patients (Intervention)
  Interventions: Radiation: low-level laser therapy (LLLT)

INTERVENTIONS:
Radiation: low-level laser therapy (LLLT) — low-level laser therapy (LLLT) with dental implants has been suggested to improve bone quality during osseointegration. Low-level laser (Gallium Aluminum Arsenide Diode [Ga-Al-As]) (wavelength: 808 nm, average power density: 50 mW, circular spot diameter:0.71 cm, spot area: 0.4cm2) in continuous mode was applied in six points in contact with peri-implant soft tissue (1.23 minutes in each point of application; dose per point 11 J) before and immediately after suturing. The application points were divided into two points in the labial region where the implant would be placed (apical and cervical); two points in the lingual region (apical and cervical); and two points in the occlusal direction. After suturing the laser protocol was repeated in the same points following the same protocol, resulting in a total dose of 66 J for each application moment (before and after implant placement).
  Arms: Low level laser therapy

SUMMARY:
This study aimed therefore to evaluate bone density (BD) and OPG levels in the peri-implant crevicular fluid (PICF) in lased controlled type II Diabetes Mellitus (T2DM) patients versus non-lased T2DM patients. 40 T2DM patients were included in this study. Implants were randomly inserted in 20 non-lased T2DM patients (Control) and 20 lased T2DM patients (Intervention). BD and OPG levels in the PICF were assessed in both groups at the follow up points.

DETAILED DESCRIPTION:
Background and objectives: Use of low-level laser therapy (LLLT) with dental implants has been suggested to improve bone quality during osseointegration. However, there is a lack of evidence about its influence on dental implants in diabetic patients. Osteoprotegrin (OPG) levels was reported as a biomarker for bone turnover to distinguish implant prognosis. This study aimed therefore to evaluate bone density (BD) and OPG levels in the peri-implant crevicular fluid (PICF) in lased controlled type II Diabetes Mellitus (T2DM) patients versus non-lased T2DM patients. Methods: 40 T2DM patients were included in this study. Implants were randomly inserted in 20 non-lased T2DM patients (Control) and 20 lased T2DM patients (Intervention). BD and OPG levels in the PICF were assessed in both groups at the follow up points.

ELIGIBILITY:
Inclusion Criteria:

* None of the participants had other major illnesses or severe diabetic complications.
* A detailed medical history of each subject was obtained according to the detailed questionnaire of the modified Cornell Medical Index [22].
* Diabetic control was measured by glycosylated hemoglobin A1c (HbA1c) of blood samples, patients had relatively stable glycemic control, as demonstrated by a difference not exceeding 1% in at least two HbA1c assays over the previous 6 months.
* Participants with partial edentulous posterior mandibular region with bone density ranging between D2 and D3, also having adjacent tooth with healthy periodontium were selected.

Exclusion Criteria:

* Any uncontrolled systemic diseases that prevent surgery for dental implant placement; (b) Need for guided bone regeneration or sinus lift for implant placement, and (c) History of radiation therapy in head and neck.
* Pregnant women, smokers and patients with para-functional habits, psychological problems or in-cooperated patients were also excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-22 (Actual)

PRIMARY OUTCOMES:
Bone density | Week 1
  Bone density was evaluated in the peri-implant crevicular fluid (PICF) in lased controlled type II Diabetes Mellitus (T2DM) patients versus non-lased T2DM patients.
Bone density | Month 1
  Bone density was evaluated in the peri-implant crevicular fluid (PICF) in lased controlled type II Diabetes Mellitus (T2DM) patients versus non-lased T2DM patients.
Bone density | Month 3
  Bone density was evaluated in the peri-implant crevicular fluid (PICF) in lased controlled type II Diabetes Mellitus (T2DM) patients versus non-lased T2DM patients.
Bone density | Month 4
  Bone density was evaluated in the peri-implant crevicular fluid (PICF) in lased controlled type II Diabetes Mellitus (T2DM) patients versus non-lased T2DM patients.
Osteoprotegrin (OPG) level | Week 1
  Osteoprotegrin (OPG) level was evaluated in the peri-implant crevicular fluid (PICF) in lased controlled type II Diabetes Mellitus (T2DM) patients versus non-lased T2DM patients.
Osteoprotegrin (OPG) level | Month 1
  Osteoprotegrin (OPG) level was evaluated in the peri-implant crevicular fluid (PICF) in lased controlled type II Diabetes Mellitus (T2DM) patients versus non-lased T2DM patients.
Osteoprotegrin (OPG) level | Month 3
  Osteoprotegrin (OPG) level was evaluated in the peri-implant crevicular fluid (PICF) in lased controlled type II Diabetes Mellitus (T2DM) patients versus non-lased T2DM patients.
Osteoprotegrin (OPG) level | Month 4
  Osteoprotegrin (OPG) level was evaluated in the peri-implant crevicular fluid (PICF) in lased controlled type II Diabetes Mellitus (T2DM) patients versus non-lased T2DM patients.

CONTACTS AND LOCATIONS:
Locations (5):
- Egypt (5):
  - Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo
  - Misr International University, Cairo
  - Misr University for Science and Technology (MUST), Cairo
  - Sinai University, El Arish
  - Delta University of Science and Technology, Gamasa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Attia MS, Elewa GM, Abdelgawad N, Ismail RM, Hassan Eid M, Ghoneim MM. The Influence of Low-Level Laser Therapy on CBCT Radiographic and Biochemical Profiles of Type II Controlled Diabetic Patients After Dental Implant Insertion: A Randomized Case-Control Study. Cureus. 2023 Mar 23;15(3):e36559. doi: 10.7759/cureus.36559. eCollection 2023 Mar. PMID 37102010